CLINICAL TRIAL: NCT06974110
Title: A Phase 1 Study of MOMA-341 as Monotherapy or Combination Therapy in Participants With Advanced or Metastatic Solid Tumors
Brief Title: Study of Orally Administered MOMA-341 in Participants With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MOMA Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOMA-341-001
Record Dates: First submitted 2025-05-02; First posted 2025-05-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Endometrial Cancer; MSI-H Cancer; Colorectal Cancer; Gastric Cancer; dMMR Cancer
Keywords: Phase 1; MOMA-341; Werner helicase; WRN; Advanced Solid Tumor; Metastatic Solid Tumor; Gastric Cancer; Colorectal Cancer; Endometrial Cancer; MSI-H Cancer; dMMR Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Endometrial Neoplasms; Colorectal Neoplasms; Stomach Neoplasms | interventions — Irinotecan; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MOMA-341 Monotherapy (Treatment Arm 1) (Experimental): MOMA-341 administered as a single agent in 21-day cycles
  Interventions: Drug: MOMA-341
- MOMA-341 in Combination with Irinotecan (Treatment Arm 2) (Experimental): MOMA-341 administered together with irinotecan in 28-day cycles
  Interventions: Drug: MOMA-341; Drug: Irinotecan
- MOMA-341 in Combination with Immunotherapy (Treatment Arm 3) (Experimental): MOMA-341 administered together with immunotherapy in 21-day cycles
  Interventions: Drug: MOMA-341; Drug: Immunotherapy

INTERVENTIONS:
Drug: MOMA-341 — MOMA-341 administered orally
Drug: Irinotecan — Irinotecan administered by IV infusion
  Arms: MOMA-341 in Combination with Irinotecan (Treatment Arm 2)
Drug: Immunotherapy — Immunotherapy administered by IV infusion
  Arms: MOMA-341 in Combination with Immunotherapy (Treatment Arm 3)

SUMMARY:
This Phase 1, multi-center, open-label, dose escalation and dose optimization study is designed to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PDx), and preliminary clinical activity of MOMA-341 administered orally as a single agent or combination therapy in patients with microsatellite instability high (MSI-H) or DNA mismatch repair deficiency (dMMR) solid tumors.

DETAILED DESCRIPTION:
MOMA-341 is a novel therapeutic agent designed to target microsatellite instability high (MSI-H) or DNA mismatch repair deficiency (dMMR) cancers by inhibiting Werner helicase. MOMA-341 is being developed as a single agent and in combination with either chemotherapy or immunotherapy in patients with certain advanced or metastatic solid tumors.

This phase 1, first-in-human, open-label study of MOMA-341 is primarily intended to evaluate the safety and tolerability of MOMA-341 when administered orally as a single agent (Treatment Arm 1), in combination with irinotecan (Treatment Arm 2), or in combination with immunotherapy (Treatment Arm 3). Each treatment arm of the study includes a dose-escalation phase, which means successive cohorts of patients will receive increasing oral doses of MOMA-341 as a single agent or in combination with irinotecan or immunotherapy to determine the presumptive optimal biologic dose(s) (OBD) in this population. The study also includes a dose-optimization phase that will enroll additional patients to support the confirmation of the OBD.

The data from this study conducted in patients with MSI-H or dMMR advanced or metastatic solid tumors, including safety, tolerability, PK/PDx findings, and antitumor activity, will form the basis for subsequent clinical development of MOMA-341 as a single-agent and in combination with irinotecan or immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Participants have unresectable advanced or metastatic solid tumors with MSI-H or dMMR alterations and histologically confirmed disease. Participants must have previously received and progressed on an anti-PD-(L)1-based regimen, unless ineligible or in a region without access to anti-PD-(L)1 therapies
3. Have at least 1 lesion at baseline (measurable or non-measurable) suitable for repeat imaging evaluation by RECIST and/or PCWG-3
4. ECOG PS ≤ 2
5. Fully recovered from clinically relevant effects of prior therapy, radiotherapy, and/or surgery **hormonal therapy allowed. Palliative radiotherapy allowed
6. Adequate organ function per local labs
7. Comply with contraception requirements
8. Written informed consent must be obtained according to local guidelines

Exclusion Criteria:

1. Known Werner Syndrome
2. Active prior or concurrent advanced-stage malignancy (some exceptions allowed including early-stage cancers)
3. Clinically relevant cardiovascular disease
4. Known CNS metastasis associated with progressive neurological symptoms (stable doses of corticosteroids allowed)
5. Known active uncontrolled infection
6. Known allergy, hypersensitivity, and/or intolerance to MOMA-341
7. Impaired GI function that may impact absorption
8. Patient is pregnant or breastfeeding
9. Known to be HIV positive, unless all of the following criteria are met:

   1. Undetectable viral load or CD4+ count ≥300 cells/μL
   2. Receiving highly active antiretroviral therapy
   3. No AIDS-related illness within the past 12 months
10. Active liver disease (some exceptions are allowed)
11. Prior or ongoing condition, therapy, or laboratory abnormality that, in the investigator's opinion, may affect safety of the patient, confound the results of the study, and/or interfere with the patients participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with AEs, dose-limiting toxicities (DLTs), serious AEs (SAEs), and/or AEs leading to discontinuation | From screening until treatment discontinuation (up to 35 months)
  To assess the safety and tolerability of MOMA-341 given as a single-agent, and in combination with irinotecan, and in combination with immunotherapy

SECONDARY OUTCOMES:
Identify the recommended phase 2 dose (RP2D) | From screening until treatment discontinuation (up to 35 months)
  Determine the RP2D of MOMA-341 as a single-agent, and in combination with irinotecan, and in combination with immunotherapy
PK parameter; area under curve (AUC) of MOMA-341 | Up to 6 weeks with sparse sampling up to 35 months
  Determine the AUC of MOMA-341 as a single-agent, and in combination with irinotecan, and in combination with immunotherapy
PK parameter; maximum concentration (Cmax) of MOMA-341 | Up to 6 weeks with sparse sampling up to 35 months
  Determine the Cmax of MOMA-341 as a single-agent, and in combination with irinotecan, and in combination with immunotherapy
PK parameter; time to maximum concentration (Tmax) of MOMA-341 | Up to 6 weeks with sparse sampling up to 35 months
  Determine the Tmax of MOMA-341 as a single-agent, and in combination with irinotecan, and in combination with immunotherapy
PK parameter; half-life (T1/2) of MOMA-341 | Up to 6 weeks with sparse sampling up to 35 months
  Determine the T1/2 of MOMA-341 as a single-agent, and in combination with irinotecan, and in combination with immunotherapy
PK parameter; plasma exposure of irinotecan | Up to 6 weeks with sparse sampling up to 35 months
  Determine the plasma exposure of irinotecan in combination with MOMA-341
Objective response rate (ORR) | Up to 35 months
  ORR is defined as the percentage of subjects with evidence of a complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 and/or Prostate Cancer Working Group-3 (PCWG-3)
Duration of response (DOR) | Up to 35 months
  DOR is defined as time from first documented PR or better to disease progression (as assessed by RECIST v1.1 and/or PCWG-3 by Investigator assessment) or death, whichever is earlier, for participants who have achieved a CR or PR
Time to response (TTR) | Up to 35 months
  TTR is defined as the period of time from the date of first dose of study treatment until the first objective documentation of a CR or PR per RECIST 1.1 and/or PCWG-3)
Progression free survival (PFS) | Up to 35 months
  PFS is defined as the time from first dose of study treatment to progressive disease or death from any cause, whichever is earlier, as assessed by RECIST 1.1 and/or PCWG-3 by investigator assessment
Disease control rate (DCR) | Up to 35 months
  DCR is defined as the proportion of subjects who achieved either CR, PR, or stable disease (SD) at the first scheduled disease assessment according to disease-specific response criteria
Overall survival (OS) | Up to 35 months
  OS is defined as the time from first dose of study treatment to the date of death, irrespective of the cause of death

CONTACTS AND LOCATIONS:
Locations (13):
- United States (7):
  - Investigative Site #128, Tampa, Florida
  - Investigative Site #120, Detroit, Michigan
  - Investigative Site #110, St Louis, Missouri
  - Investigative Site #131, Raleigh, North Carolina
  - Investigative Site #121, Portland, Oregon
  - Investigative Site #127, Dallas, Texas
  - Investigative Site #129, Houston, Texas
- Australia (6):
  - Investigative Site #122, Sydney, New South Wales
  - Investigative Site #123, Westmead, New South Wales
  - Investigative Site #124, Woolloongabba, Queensland
  - Investigative Site #125, Adelaide, South Australia
  - Investigative Site #126, Clayton, Victoria
  - Investigative Site #119, Perth, Western Australia